CLINICAL TRIAL: NCT04870970
Title: The Effect of Tobacco Products on Wound Healing
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00006048
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Smoking; Tobacco Use; Tobacco Smoking
Keywords: Wound healing
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A separate electronic consent form will be used to allow the use of specimens collected (both blood and tissue) for genetic research. Participants can decline the use of their specimens for genetic research but may not be able to participate in the study. The study coordinator will keep a log through REDCap of which participants declined the use of their samples for genetic research to ensure those samples will not be used for genetic research. Participants will also have the option to allow the future use of their de-identified specimens collected for general research, including genetic purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tobacco Users: Participants in this group use some form of tobacco.
- Non-Tobacco Users: Participants in this group do not use tobacco products.

SUMMARY:
The purpose of this study is to evaluate the effect of various tobacco products (including but not limited to combustible cigarettes, medicinal nicotine, electronic cigarettes, and smokeless tobacco) on cutaneous wound healing. There will also be a non- smoking control group. This study will be designed as a pilot study. The majority of individuals will be recruited from ongoing studies at the University of Minnesota - Tobacco Research Programs.

DETAILED DESCRIPTION:
Participants will be recruited from ongoing studies will some recruitment of tobacco users and non-smoking controls outside of ongoing studies. In this prospective, cohort study of various tobacco users and non-smokers, a punch biopsy model of wound healing will be used to determine the effects of various tobacco products on inflammatory response and oxidative stress response to wounding:

1. Clinical wound inflammation as assessed by:

   1. Thermography,
   2. Clinical assessment,
   3. Laser Doppler Technologies,
   4. Transcutaneous oxygen assessment
2. Biological wound inflammation as assessed by:

   1. Cytokine profiles,
   2. Histology,
   3. Genetic assessment,
   4. Epigenetic evaluation
3. Systemic inflammation as assessed by:

   1. Biomarkers,
   2. Cell counts

ELIGIBILITY:
1. For participants NOT enrolled in an active Tobacco Research Programs study:

   Inclusion criteria:
   * In good physical health with no unstable or serious medical conditions as determined by the licensed medical professional;
   * In stable and good mental health (i.e. not currently, within the past 6 months, experiencing unstable or untreated psychiatric diagnosis, including substance abuse) as determined by the licensed medical professional;

   The remaining inclusion criteria is different depending on the type of tobacco product the individual uses:

   A) Non Smokers
   * Has consumed less than 100 cigarettes in his or her lifetime.
   * Combustible Tobacco Users
   * History of at least 5 years smoking
   * Smokers will have exclusively smoked at least 5 cigarettes per day for a minimum of 4 days per week for the past year

   B) E-Cigarette Users
   * Have not smoked cigarettes in the last month
   * Has exclusively used e-cigarettes for at least 3 months
   * Has at least 5 instances of using an e cigarettes per day for a minimum of 4 days per week

   C) Medicinal Nicotine Users
   * Have not smoked cigarettes in the last month
   * Has at least 5 instances of using medicinal nicotine per day for a minimum of 4 days per week

   D) Smokeless Tobacco Users

   - Have not smoked cigarettes in the last month

   - Has at least 5 instances of using smokeless tobacco per day for a minimum of 4 days per week

   E) Combustible Tobacco and E-Cigarette Dual Users
   * Has used a combination of combustible tobacco products and e-cigarettes for the past month.
   * Has at least 5 instances of using a combination of combustible tobacco and e-cigarettes per day for a minimum of 4 days per week

   F) Combustible Tobacco and Medicinal Nicotine Dual Users
   * Has used a combinations of combustible tobacco products and e-cigarettes for the past month.
   * Has at least 5 instances of using a combination of combustible tobacco and medicinal nicotine per day for a minimum of 4 days per week

   Exclusion Criteria:
   * Any tattoos on the medial upper arm (note that one medial upper arm can have a tattoo, but at least one side does not have a tattoo).
   * History of delayed wound healing.
   * Intention to quit normal tobacco product use in the next three months.
   * Excessive drinking (more than 21 alcoholic drinks per week)
   * Taking exclusionary medications (including anti-inflammatory agents) unstable dosing of medications, or unstable control of symptoms for ongoing medical conditions (medications or conditions that would impact biomarkers or patient safety to be determined by the licensed medical professional at each site).
   * Active infection (e.g., influenza, cold, respiratory infection, sinus infection), admission to study will be delayed pending improved health;
   * Additional exclusion criteria for those undergoing the additional Laser Doppler Technologies
   * Individuals with extremely sensitive skin that may feel the 45 degrees Celsius is too warm
   * Pregnant or breastfeeding or plans to become pregnant
2. For participants enrolled in an active Tobacco Research Programs study:

   Inclusion Criteria:

   Concurrent enrollment in one of the following studies (if the study is registered with clinicaltrials.gov, please click the link to see inclusion/exclusion criteria):

   A) Impact of Very Low Nicotine Content Cigarettes in a Complex Marketplace - https://clinicaltrials.gov/ct2/show/NCT03272685 B) Clinical trial to assess the removal of filter ventilation on smoking behavior and biomarkers - https://clinicaltrials.gov/ct2/show/NCT03637972 C) e-Cigarettes: Formaldehyde DNA Adducts, Oxidative Damage, and Potential Toxicity and Carcinogenesis - https://clinicaltrials.gov/ct2/show/NCT03284632 D) Methodology and Development of Tobacco Related Biomarkers, part of "Metabolism of Carcinogenic Tobacco-Specific Nitrosamines" Inclusion Criteria - Generally good physical and mental health as evidenced by a medical history with no unstable medical conditions and study physician approval.

   Exclusion Criteria

   - Pregnant or breastfeeding or plans to become pregnant
   * Regular use of other tobacco or smoked products (e.g., cigars, pipes, smokeless tobacco, marijuana) in past 6 months;
   * Active infection (e.g., influenza, cold, respiratory infection, sinus infection), admission to study will be delayed pending improved health;
   * Unstable medical or psychiatric condition

   SMOKERS

   Inclusion:

   - Currently smoking at least 10 cigarettes per day;

   - History of at least 5 years smoking;

   - Stable smoking pattern for the past 1 year (<50% change in brand or number of cigarettes smoked).

   FORMER SMOKERS

   Inclusion:
   * History of smoking at least 10 cigarettes per day;
   * Quitting over 1 year ago

   NEVER SMOKERS

   Exclusion:

   - Smoking more than 100 cigarettes in their lifetime

   NICOTINE REPLACEMENT USERS

   - Inclusion/Exclusion dependent on intended sample use

   E-CIGARETTE USERS (Addendum study) - Inclusion/Exclusion dependent on intended sample use

   SMOKELESS TOBACCO USERS (Addendum study)

   - Inclusion/Exclusion dependent on intended sample use

   E) Clinical Trial of Watercress in Detoxification of Environmental Toxicants and Carcinogens - https://clinicaltrials.gov/ct2/show/NCT03978117 F) Metabolism of Deuterated NNN in Smokeless Tobacco Users - https://clinicaltrials.gov/ct2/show/NCT02414477 G) Biomarkers of Exposure and Effect in SREC Users - https://clinicaltrials.gov/ct2/show/NCT04003805 H) Nornicotine in Smokeless Tobacco as a Precursor for Carcinogen Exposure - https://www.clinicaltrials.gov/ct2/show/NCT03998735 I) Phase 1 Trial of Indole-3-Carbinol and Silibinin Inclusion Criteria

   - Current smoker of ≥ 8 cigarettes per day for at least the last 6 months by self-report

   Adequate blood counts, and adequate liver and kidney function defined as follows:

<!-- -->

1. Hemoglobin ≥ 9 g/dL for women, ≥ 10 g/dL for men
2. Platelet count ≥ 100 x 109/L
3. Total bilirubin ≤ Institutional upper limit of normal (≤ 1.3 mg/dL for UMMC)
4. ALT ≤ 1.5 times institutional upper limit of normal
5. Creatinine ≤ 1.4 g/dL and estimated GFR ≥ 80 mL/min/1.7m2

   Exclusion Criteria

   - Daily proton pump inhibitor, H2-blocker (i.e., ranitidine, famotidine), and/or calcium carbonate use

   - History of gastric bypass surgery, gastric banding, bowel resection, malabsorption syndromes such as celiac sprue or pancreatic insufficiency, or other conditions that may affect gastric or intestinal absorption of nutrients

   - Use of tobacco products other than cigarettes (i.e. snuff, snuz, smokeless tobacco, cigars, pipes), within 7 days of study registration
   * Major or chronic medical disease, including heart disease, poorly controlled diabetes, etc., to be adjudicated by the principal investigator
   * Known active malignancy
   * History of aerodigestive malignancies
   * Pregnancy, intension to become pregnant within 3 months of study registration, or lactation. Participants of childbearing potential must have a negative urine pregnancy test within 14 days of starting the assigned intervention
   * Antibiotic use within 2 months of study registration by self-report
   * History of respiratory tract cancer
   * Known allergy to I3C, Sil, or its components
   * Psychiatric and/or social situations that would potentially limit compliance with study requirements

   Exclusion Criteria:

   - Any tattoos on the medial upper arm (note that one medial upper arm can have a tattoo, but at least one side does not have a tattoo).

   - History of delayed wound healing.
   * Additional exclusion criteria for those undergoing the additional Laser Doppler Technologies
   * Individuals with extremely sensitive skin that may feel the 45 degrees Celsius is too warm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must be enrolled in an ongoing study for participation in this sub-study or meet the inclusion/exclusion criteria for participants not enrolled in an active study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Cutaneous temperature | approximately 7 days
  Cutaneous temperature is measured using in infrared thermographic camera (FLIR T460 Infrared Thermal Imaging Camera, FLIR Systems, Inc., Wilsonville, OR). Images will be analyzed using a camera-specific software (FLIR Tools) that interrogates cutaneous temperature points of the image. The units are software-determined, arbitrary units that are standardized within the FLIR imaging system but do not correspond to standard units of measure.
Cutaneous perfusion | approximately 7 days
  Cutaneous perfusion is measured using Laser Doppler Technologies (PeriFlux 6000, Perimed AB, Stockholm, Sweden). Tissue oxygenation is measured in the capillaries only. Perfusion is measured in arbitrary system defined "perfusion units."
Cutaneous oxygenation | approximately 7 days
  Cutaneous oxygenation is measured using Laser Doppler Technologies (PeriFlux 6000, Perimed AB, Stockholm, Sweden). Tissue oxygenation is measured in the capillaries only. Oxygenation is measured in mmHg.
Immunohistochemistry - markers of inflammation | approximately 7 days
  CD31 and C68 are stained via standard immunohistochemistry methods on punch biopsied specimens. Unit of measure is cell count.
Biological Wound Inflammation | approximately 7 days
  IL-1b, 6 and 10 are measured using standard immunoassays and reported in units of pg/ml. These cytokines will be measured in both the skin and blood.
Tumor necrosis factor (TNF)-alpha | approximately 7 days
  TNF-alpha is measured using standard immunoassays and reported in units of pg/ml. This cytokine will be measured in both the skin and blood.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States